CLINICAL TRIAL: NCT03743935
Title: Primary Prevention ICD Implantation in STEMI With Severe Left Ventricular Dysfunction : Input of Early Cardiac MRI in Order to Predict Left Ventricular Recovery
Brief Title: Use of Cardiac MRI in Early Stages of STEMI to Predict Left Ventricular Function Recovery and ICD Implantation
Acronym: STEMI-MR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Société Française de Cardiologie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL18_0183; 2018-A02470-55 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-11-09; First posted 2018-11-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2022-02

CONDITIONS: Acute STEMI; Severe Left Ventricular Systolic Dysfunction (Disorder)
Keywords: STEMI; MRI; ICD; Sudden death
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ventricular Dysfunction, Left; Death, Sudden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Early cardiac MRI post-STEMI (Experimental): Early stages post-STEMI (within the first 5 days)
  Interventions: Other: Gadolinium-enhanced cardiac MRI

INTERVENTIONS:
Other: Gadolinium-enhanced cardiac MRI — Gadolinium-enhanced cardiac MRI during the 1st days post-STEMI with specific sequences including extra-cellular volume measurement

SUMMARY:
Patients presenting with STEMI and late revascularization can suffer from severe left ventricular dysfunction. Midterm and longterm mortality can be determined by the risk of fatal ventricular arrythmias. For this specific population, ESC guidelines currently recommend a waiting period of up to 40 days after a STEMI with severe left ventricular dysfunction before considering ICD implantation for primary prevention of sudden death.This delay is allocated to judge left ventricular recovery.

This study aims to see whether early cardiac MRI with specific sequences can help predict which patients will most probably not recover their left ventricular function and benefit from earlier ICD implantation.

DETAILED DESCRIPTION:
ST segment elevation myocardial infarction represent 120 000 annual cases in France. Although its mortality has been drastically reduced by primary percutaneous coronary angioplasty (PCI), its midterm and longterm outcome in patients presenting initially with severe left ventricular (LV) dysfunction depends on the risks of heart failure and sudden death by malignant ventricular arrhythmias.

Many clinical studies such as MADIT I and II, MUSTT and DINAMIT have participated in defining which patients should benefit from ICD implantation. These studies were based on evaluation of the LV ejection fraction (LVEF) and of the risk of arrhythmia (by electrophysiology or holter recordings).

However, ESC Guidelines recommend a mandatory waiting period of 40 days post-PCI to reevaluate LVEF before confirming the need for ICD implantation (LVEF < 35%). Therefore, patients are at risk of sudden cardiac death (SCD). during this period.

The investigators sought to determine whether specific cardiac MRI sequences could help predict which patients would eventually recover from their LV dysfunction and therefore reduce the risk of SCD by implanting ICD earlier than recommended.

Patients presenting at our Cardiac ICU with STEMI and severe LV dysfunction (LVEF < 35%), not indicated to coronary artery bypass surgery (CABG) and free from initial cardiac arrest or severe ventricular arrhythmias, will be included. They will undergo a gadolinium-enhanced cardiac MRI during the 1st days of hospitalization with specific sequences to determine myocardial zones at risk of non-recovery.

Initial assessment will also include thorough clinical examination with NYHA class, trans-thoracic echocardiography and blood works to evaluate renal function, inflammation, signs of heart failyre (BNP and troponin). Patients will be equipped with Lifevests for 6 weeks and followed-up with the same criteria.

Ratio of final ICD implantation will then be compared to the MRI criterion to determine whether LV recovery could have been predicted.

ELIGIBILITY:
Inclusion Criteria:

* Acute STEMI within 5 last days with LVEF < 35%
* 18-80 years old
* Admitted to the Cardiac ICU
* Consent form

Exclusion Criteria:

* CABG surgery indicated
* Contra-indications to MRI
* ICD or PPM in place
* Follow-up compromised

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Mesure of zones of delayed myocardial transmural enhancement and no-reflow | 40 days
  Defining the area at risk with Cardiac MRI
Mesure of ejection fraction and regional wall motion and thickening | 40 days
  Defining the area at risk with Cardiac MRI
Mesure of extracellular volume | 40 days
  Defining the area at risk with Cardiac MRI

SECONDARY OUTCOMES:
Number of CVD events | 40 days
  Occurrence of major adverse cardiac events
Number of admission to the hospital for heart failure event | 40 days
  Occurrence of heart failure events
Number of ischemic cardiovascular events | 40 days
  Occurrence of major adverse cardiac events
Number of cardiac death | 40 days
  Occurrence of major adverse cardiac events

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tangerman A. Determination of volatile sulphur compounds in air at the parts per trillion level by Tenax trapping and gas chromatography. J Chromatogr. 1986 Sep 24;366:205-16. doi: 10.1016/s0021-9673(01)93468-5. PMID 3782318
- [Background] Perazzolo Marra M, Lima JA, Iliceto S. MRI in acute myocardial infarction. Eur Heart J. 2011 Feb;32(3):284-93. doi: 10.1093/eurheartj/ehq409. Epub 2010 Nov 25. PMID 21112897
- [Background] Schelbert EB, Wong TC. Imaging the area at risk in myocardial infarction with cardiovascular magnetic resonance. J Am Heart Assoc. 2014 Aug 21;3(4):e001253. doi: 10.1161/JAHA.114.001253. No abstract available. PMID 25146709
- [Background] Haaf P, Garg P, Messroghli DR, Broadbent DA, Greenwood JP, Plein S. Cardiac T1 Mapping and Extracellular Volume (ECV) in clinical practice: a comprehensive review. J Cardiovasc Magn Reson. 2016 Nov 30;18(1):89. doi: 10.1186/s12968-016-0308-4. PMID 27899132
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621